CLINICAL TRIAL: NCT06382844
Title: Design, Development, and Validation of Novel "Next Generation Flow" Approaches for Rapid, Specific, Sensitive, and Reproducible Detection of Tumor Cells in Cutaneous T-cell Lymphoma.
Brief Title: Novel Flow-cytometry Approaches to Improve the Detection of Tumor Cells in CTCL
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: PI23/00486; PI2023 08 1416 (Registry Identifier: Ethics Committee for Drug Research of the Salamanca Health Area)
Record Dates: First submitted 2024-04-20; First posted 2024-04-24 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cutaneous T-Cell Lymphoma
Keywords: Lymphoma; T Cell; Cutaneous; Flow cytometry; Mycosis fungoides; Sézary syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma; Mycosis Fungoides; Sezary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cutaneous T-cell lymphoma: Patients with cutaneous T-cell lymphoma
  Interventions: Diagnostic Test: Detection and quantitation of (blood) tumor cells in patients with mycosis fungoides (MF) / Sézary syndrome (SS).
- Control group 1: patients with benign/reactive erythroderma
  Interventions: Diagnostic Test: Detection and quantitation of (blood) tumor cells in patients with mycosis fungoides (MF) / Sézary syndrome (SS).
- Control group 2: patients with systemic inflammatory processes regardless of whether they have cutaneous involvement
  Interventions: Diagnostic Test: Detection and quantitation of (blood) tumor cells in patients with mycosis fungoides (MF) / Sézary syndrome (SS).
- Control group 3: healthy adult subjects, age- and sex-matched with patients
  Interventions: Diagnostic Test: Detection and quantitation of (blood) tumor cells in patients with mycosis fungoides (MF) / Sézary syndrome (SS).

INTERVENTIONS:
Diagnostic Test: Detection and quantitation of (blood) tumor cells in patients with mycosis fungoides (MF) / Sézary syndrome (SS). — Specific, sensitive, and reproducible (blood) detection and quantitation of tumor cells in patients with mycosis fungoides (MF) / Sézary syndrome (SS)

SUMMARY:
Identification and quantitation of circulating tumor cells in patients with cutaneous T-cell lymphoma -mycosis fungoides (MF)/Sézary syndrome (SS)- are required for diagnosis and precising the actual staging and response to treatment. The current flow cytometry techniques used in clinical laboratories do not correctly allow to compare results in a clinical setting. Furthermore, now we know that the phenotype of tumor cells partially overlaps with that of normal TCD4+ cells, and it is rather heterogeneous. The GENERAL OBJECTIVE of this project is to apply flow-cytometry standardized strategies for rapid, specific, sensitive, and reproducible detection and quantitation of tumor cells in patients with MF/SS. For this purpose, in the first phase of the project we will design an optimal combination of markers to detect tumor cells by spectral flow-cytometry, and then the specificity and analytical sensitivity of the new combination/procedure will be assessed in blood samples -to be later applied to skin samples-, and finally reference databases will be created for the automatic analysis of cytometry data. In a second phase of the project, the developed method will be validated in a multicenter manner, through the demonstration of its practical applicability and clinical utility (speed and precision) in blood samples (and skin, where appropriate) for diagnosis, staging, and treatment monitoring. In parallel, the tumor microenvironment (residual normal immune system) will be explored -by applying the panel designed in the first phase together with additional immune-monitoring panels by flow cytometry-, and its relationship with clinical-biological heterogeneity of the tumor will be analyzed. In the two phases of the project, cytometry data will be compared with the gold standard approach to identify tumor T cells (through the identification of clonal rearrangement by PCR and/or NGS, performed on cell populations previously sorted by flow cytometry).

DETAILED DESCRIPTION:
Primary cutaneous lymphomas are a group of tumors derived from lymphocytes (mostly T lymphocytes) that primarily affect the skin (such as mycosis fungoides, MF), although they can spread beyond the skin in more advanced stages - for example, to the blood - or may already be disseminated initially, as is the case with Sézary syndrome (SS), a tumor with very aggressive behavior from the beginning, which by definition already has blood dissemination at diagnosis. They are very rare tumors and difficult to diagnose because often the skin lesions are indistinguishable from benign processes (the latter much more common than cutaneous lymphomas). For this reason, it is not uncommon for the diagnosis to be delayed, with the consequent negative impact on the patient's prognosis if it is a tumor. Currently, the diagnosis of blood dissemination (the amount of which is also essential because it impacts the prognosis, the worse the higher tumor burden in the blood) is performed by flow cytometry, which has replaced conventional morphology. However, the flow cytometry techniques currently used in most clinical laboratories are not standardized among different centers, and therefore the comparability of the results (even over time, in the same center) and their use in the clinical settings is difficult.

In this project, the investigators HYPOTHESIZE that the application of novel "next-generation flow" strategies proposed by the international collaborative group EuroFlow (to which the applicant of this proposal belongs) would improve the detection of circulating tumor cells in patients with cutaneous T-cell lymphoma, which would allow improving the clinical management of the patients. Therefore, in this project, the aim as a GENERAL OBJECTIVE to apply standardized strategies of next-generation flow cytometry developed by the EuroFlow Consortium for the rapid, specific, sensitive, and reproducible detection and quantification of tumor cells in patients with MF/SS, through: i) the application of standardized sample staining procedures with antibody panels designed after previous rounds of testing, which would allow distinguishing tumor T lymphocytes from normal T cells (specificity); ii) adapting the technique to analyze a large number of cells, in order to achieve a high sensitivity of detection, also crucial for a more precise monitoring of residual disease in blood after treatment with the new therapies available in cutaneous T-cell lymphomas; and iii) development of automatic analysis strategies of cytometry data, so that the results do not depend on the personal experience of the cytometrist.

IMPACT. The availability of a new standardized flow cytometry strategy for sensitive and specific detection (and quantification) of circulating tumor cells in blood (and skin) of patients with cutaneous T-cell lymphoma will provide an essential tool to support dermo-hematological diagnosis, with the possibility of translating to routine diagnosis in the very short term after the completion of the project, for its application in hospitals that have a Cytometry/Immunopathology Laboratory, with the aim of: i) Making an early and accurate (differential) diagnosis between lymphoma - benign lesion in patients with skin lesions; ii) Detecting tumor cells in blood with greater sensitivity than conventional methods, to more precisely establish blood dissemination of a primary cutaneous T-cell lymphoma, and to assess the response to current treatments in a more reliable and sensitive way

ELIGIBILITY:
Inclusion Criteria:

* Patients with cutaneous T-cell lymphoma
* Over 18 years old
* Sign the informed consent

Exclusion Criteria:

* Under 18 years old
* Do not sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases of cutaneous lymphoma/reactive erythroderma will be recruited from the routine clinical practice of the Cutaneous T-Cell Lymphoma Monographic Clinic at the University Hospital of Salamanca, which is conducted in a multidisciplinary manner under the responsibility of the Dermatology and Hematology services, involving two members of the research team (ECA and MLP). Diagnosis will be made according to the current criteria of the EORTC-OMS; patients will be included both at diagnosis and at any other stage of the tumor during follow-up
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Optimizing Marker Combination for Specific Identification and Quantification of Sézary Cells using Spectral Flow Cytometry | 18 months
  Designing an optimal marker combination for the specific identification and quantification of Sézary cells (particularly in blood) using spectral flow cytometry, enabling their discrimination from normal/reactive TCD4+ cells, and including markers for T-cell identification, T-cell maturation, aberrant markers, and markers to assess T-cell clonality

CONTACTS AND LOCATIONS:
Overall Officials: Julia M Almeida Parra, Prof., Principal Investigator — Instituto de Investigación Biomédica de Salamanca
Locations (1):
- Instituto de Investigación Biomédica de Salamanca (IBSAL), Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided